CLINICAL TRIAL: NCT05085912
Title: A Randomized Control Study of Driver Ablation of Persistent Atrial Fibrillation With Severe Atrial Fibrosis: a Chinese Registry Study.
Brief Title: Driver Ablation of Persistent Atrial Fibrillation With Severe Atrial Fibrosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospita, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAAF
Record Dates: First submitted 2021-10-05; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; severe atrial fibrosis; driver ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation
- Group B (Active Comparator): Circumferential pulmonary vein isolation + linear ablation + posterior wall box isolation
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + posterior wall box isolation
- Group C (Active Comparator): Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion

INTERVENTIONS:
Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with bi-atrial mapping and driver ablation.
  Arms: Group A
Procedure: Circumferential pulmonary vein isolation + linear ablation + posterior wall box isolation — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with posterior wall box isolation.
  Arms: Group B
Procedure: Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with vein of Marshall ethanol infusion.
  Arms: Group C

SUMMARY:
This is an open label, randomized parallel control clinical trial, to demonstrate the role of driver mechanism in maintenance substrate of persistent atrial fibrillation with severe atrial fibrosis, and evaluate the clinical outcomes of driver mapping and ablation strategy in patients with persistent atrial fibrillation with severe atrial fibrosis.

DETAILED DESCRIPTION:
This is an open label, randomized parallel control clinical trial. Patients with persistent atrial fibrillation with severe atrial fibrosis are 1:1:1 randomized into group A (circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation), group B (circumferential pulmonary vein isolation + linear ablation + posterior wall box isolation) and group C (circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion). Postoperative recurrence rate and other indicators are analyzed to demonstrate the role of driver mechanism in maintenance substrate of persistent atrial fibrillation with severe atrial fibrosis and evaluate the clinical outcomes of driver mapping and ablation strategy in patients with persistent atrial fibrillation with severe atrial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Persistent AF with severe atrial fibrosis;
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug.

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease;
3. With myocardial infarction or stroke within 6 months of screening;
4. With Significant congenital heart disease;
5. Ejection fraction was <40% measured by echocardiography;
6. Allergic to contrast media;
7. Contraindication to anticoagulation medications;
8. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
9. Left atrial (LA) thrombus;
10. Having any contraindication to right or left sided heart catheterization; 11. Previous atrial fibrillation ablation;

12. Presence of an implanted cardioverter-defibrillator; 13. Previous history of cardiac surgery; 14. Poor general health; 15. Life expectancy less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | up to 12 months after ablation
  AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration
Intraoperative AF termination rate | through ablation completion, an average of 3 hours
  AF termination is defined as conversion to sinus rhythm or stable AFL/AT.

SECONDARY OUTCOMES:
Postoperative AF recurrence rate | up to 12 months after ablation
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration
Postoperative AFL/AT rate | up to 12 months after ablation
  occurrence of AFL/AT is defined as presence of documented AFL/AT episodes of 30 seconds or longer duration
Incidence of complications | up to 12 months after ablation
  death, atrioesophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, diaphragmatic paralysis, pneumothorax, heart block, pulmonary vein stenosis, pulmonary edema, pericarditis and major vascular access complication or bleeding
Changes in the diameter of the left atrium | up to 12 months after ablation
  Changes in the diameter of the left atrium
Changes in the left ventricular ejection fraction | up to 12 months after ablation
  Changes in the left ventricular ejection fraction